CLINICAL TRIAL: NCT01415336
Title: AX (Doxorubicin, Capecitabine) Versus AC (Doxorubicin, Cyclophosphamide) as Adjuvant Treatment for Node-Negative Breast Cancer
Brief Title: AX Versus AC as Adjuvant Treatment for Node-Negative Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Qiang Sun, the department of breast surgery of PUMCH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-Breast- AX
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AC protocol; Doxorubicin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC (Active Comparator): doxorubicin 60 mg/m², iv, day 1 Cyclophosphamide 600 mg/m², iv, day 1 every 3 weeks for 4 cycles
  Interventions: Drug: Doxorubicin, Cyclophosphamide
- AX (Experimental): doxorubicin 60 mg/m², iv, day 1 capecitabine 950 mg/m2, twice a day, via oral intake, day 1 to day 14 every 3 weeks for 4 cycles
  Interventions: Drug: doxorubicin, Capecitabine

INTERVENTIONS:
Drug: Doxorubicin, Cyclophosphamide — doxorubicin 60 mg/m², iv, day 1; Cyclophosphamide 600 mg/m², iv, day 1; every 3 weeks for 4 cycles
  Arms: AC
Drug: doxorubicin, Capecitabine — doxorubicin 60 mg/m², iv, day 1; capecitabine 950 mg/m2, twice a day, via oral intake, day 1 to day 14; every 3 weeks for 4 cycles
  Arms: AX

SUMMARY:
Capecitabine has shown high efficacy in metastatic and adjuvant settings. This is a prospective, randomised trial, to compare the efficacy and safety profiles of capecitabine-containing regimen with non- capecitabine-containing adjuvant chemotherapy regimens for node negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnosis of operable invasive adenocarcinoma of the breast Tumours must be node negative. Time window between surgery and study randomization must be less than 60 days.
* Surgery must consist of mastectomy or conservative surgery with axillary lymph node dissection. Margins free of disease and ductal carcinomas in situ (DCIS) are required. Lobular carcinoma is not considered a positive margin.
* Status of hormone receptors in primary tumour. Results must be available before the end of adjuvant chemotherapy.
* Patients must not present evidence of metastatic disease. Status of HER2 in primary tumour, known before randomization.
* Age >= 18 and <= 70 years old.
* Performance status (Karnofsky index) >= 70.
* Normal electrocardiogram (EKG) in the 12 weeks prior to randomization. If needed, normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF).
* Laboratory results (within 14 days prior to randomization):

  * Hematology: neutrophils >= 1.5 x 10^9/l; platelets >= 100 x 10^9/l; hemoglobin >= 10 mg/dl;
  * Hepatic function: total bilirubin <= 1 upper normal limit (UNL); SGOT and SGPT <= 2.5 UNL; alkaline phosphatase <= 2.5 UNL. If values of SGOT and SGPT > 1.5 UNL are associated to alkaline phosphatase > 2.5 UNL, patient is not eligible;
  * Renal function: creatinine <= 175 mmol/l (2 mg/dl); creatinine clearance >= 60 ml/min;
* Complete stage workup during the 12 weeks prior to randomization (mammograms are allowed within a 20 week window). All patients must have a bilateral mammogram, thorax x-ray, abdominal echography and/or computed tomography (CT)-scan. If bone pain, and/or alkaline phosphatase elevation, a bone scintigraphy is mandatory. This test is recommended for all patients. Other tests: as clinically indicated.
* Patients able to comply with treatment and study follow-up.
* Negative pregnancy test done in the 14 prior days to randomization.

Exclusion Criteria:

* Prior systemic therapy for breast cancer.
* Prior therapy with anthracyclines or capecitabine for any malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments.
* Any M1 tumour.
* Lymph node positive breast cancer.
* Pre-existing grade >= 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria version 2.0 [NCI CTC v-2.0]).
* Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled HA or high risk arrhythmias.
* History of neurological or psychiatric disorders, which could preclude the patients from free informed consent.
* Active uncontrolled infection.
* Active peptic ulcer; unstable diabetes mellitus.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumour curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Chronic treatment with corticosteroids.
* Contraindications for corticosteroid administration.
* Concomitant treatment with raloxifene, tamoxifen or other selective estrogen receptor modulators (SERMs), either for osteoporosis treatment or for prevention. These treatments must stop before randomisation.
* Concomitant treatment with other investigational products; participation in other clinical trials with a non-marketed drug in the 20 previous days before randomization.
* Concomitant treatment with another therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Adverse event rate (CTCAE v. 3.0) | 3 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, Master, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241